CLINICAL TRIAL: NCT04173013
Title: Expanded Access Program Using Uromune for Patients With Recurrent Urinary Tract Infections (rUTI)
Status: No longer available | Type: Expanded Access
Sponsor: Impatients N.V. trading as myTomorrows (Industry)
Collaborators: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-UROMUNEINM-EU
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Urinary Tract Infections; Chronic Urinary Tract Infection; Recurrent Urinary Tract Infection; Urinary Tract Infection Bacterial; Bladder Infection
MeSH Terms: conditions — Urinary Tract Infections; Cystitis | interventions — uromune

INTERVENTIONS:
Biological: Uromune — 2 sprays of solution once daily for a total of 3 months.
  Other Names: MV140

SUMMARY:
An Expanded Access Program for UROMUNE® for patients suffering from recurrent/chronic urinary tract infections of diverse etiology. This is for individuals for whom antibiotic therapy has failed, but of consideration in all cases, taking into account antibiotic-induced adverse reactions and increasing antibiotic resistance.

DETAILED DESCRIPTION:
UROMUNE® is a mucosal immunotherapy indicated for the prevention of urinary tract infections caused by different pathogens. It works by stimulating the immune system, thus increasing the resistance against recurrent infections. The active substances are 4 inactivated and selected bacterial strains:

* Klebsiella pneumoniae 25%
* Escherichia coli 25%
* Enterococcus faecalis 25%
* Proteus vulgaris 25%

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering recurrent urinary tract infections of diverse etiology.

Exclusion Criteria:

* Individuals being allergic to any of the ingredients of UROMUNE®.
* Pregnancy and breast feeding. There are neither specific studies nor a formal contraindication, the physician should value benefits/risk.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (15):
- Belgium, Brussels, Belgium
- Czech Republic, Prague, Czechia
- Denmark, Copenhagen, Denmark
- Finland, Helsinki, Finland
- France, Paris, France
- Germany, Berlin, Germany
- Luxembourg, Luxembourg, Luxembourg
- The Netherlands, Amsterdam, Netherlands
- Norway, Oslo, Norway
- Romania, Bucharest, Romania
- Serbia, Belgrade, Serbia
- Slovakia, Bratislava, Slovakia
- Slovenia, Ljubljana, Slovenia
- Sweden, Stockholm, Sweden
- Turkey, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Benito-Villalvilla C, Cirauqui C, Diez-Rivero CM, Casanovas M, Subiza JL, Palomares O. MV140, a sublingual polyvalent bacterial preparation to treat recurrent urinary tract infections, licenses human dendritic cells for generating Th1, Th17, and IL-10 responses via Syk and MyD88. Mucosal Immunol. 2017 Jul;10(4):924-935. doi: 10.1038/mi.2016.112. Epub 2016 Dec 14. PMID 27966556
- [Result] Yang B, Foley S. First experience in the UK of treating women with recurrent urinary tract infections with the bacterial vaccine Uromune(R). BJU Int. 2018 Feb;121(2):289-292. doi: 10.1111/bju.14067. Epub 2017 Nov 23. PMID 29171130
- [Result] Lorenzo-Gomez MF, Padilla-Fernandez B, Garcia-Cenador MB, Virseda-Rodriguez AJ, Martin-Garcia I, Sanchez-Escudero A, Vicente-Arroyo MJ, Miron-Canelo JA. Comparison of sublingual therapeutic vaccine with antibiotics for the prophylaxis of recurrent urinary tract infections. Front Cell Infect Microbiol. 2015 Jun 3;5:50. doi: 10.3389/fcimb.2015.00050. eCollection 2015. PMID 26090341
- [Result] Ramirez Sevilla C, Gomez Lanza E, Manzanera JL, Martin JAR, Sanz MAB. Active immunoprophyilaxis with uromune(R) decreases the recurrence of urinary tract infections at three and six months after treatment without relevant secondary effects. BMC Infect Dis. 2019 Oct 28;19(1):901. doi: 10.1186/s12879-019-4541-y. PMID 31660885